CLINICAL TRIAL: NCT03816319
Title: A Phase 1 Study of TAK-243 for Relapsed or Refractory Acute Myeloid Leukemia or Myelodysplastic Syndromes With Increased Blasts
Brief Title: TAK-243 in Treating Patients With Relapsed or Refractory Acute Myeloid Leukemia or Myelodysplastic Syndromes With Increased Blasts
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2019-00238; NCI-2019-00238 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 10237 (Other: University Health Network Princess Margaret Cancer Center LAO); 10237 (Other: CTEP); UM1CA186644 (NIH)
Record Dates: First submitted 2019-01-24; First posted 2019-01-25 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-01

CONDITIONS: Myelodysplastic Syndrome With Excess Blasts; Recurrent Acute Myeloid Leukemia; Recurrent Myelodysplastic Syndrome; Recurrent Myelodysplastic Syndrome/Acute Myeloid Leukemia; Refractory Acute Myeloid Leukemia; Refractory Myelodysplastic Syndrome; Refractory Myelodysplastic Syndrome/Acute Myeloid Leukemia
MeSH Terms: conditions — Anemia, Refractory, with Excess of Blasts; Leukemia, Myeloid, Acute; Myelodysplastic Syndromes | interventions — Specimen Handling; Biopsy; TAK-243

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (TAK-243) (Experimental): Patients receive TAK-243 IV over 30 minutes on days 1, 4, 8, and 11 of each cycle. Cycles repeats every 21 days for up to 12 months in the absence of disease progression or unacceptable toxicity. Patients undergo urine sample collection, bone marrow aspiration and bone marrow biopsy, MUGA and ECHO during screening and on study, and blood sample collection throughout the trial.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy; Procedure: Echocardiography Test; Procedure: Multigated Acquisition Scan; Drug: UAE Inhibitor TAK-243

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo urine and blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Bone Marrow Aspiration — Undergo bone marrow aspiration
Procedure: Bone Marrow Biopsy — Undergo bone marrow biopsy
  Other Names: Biopsy of Bone Marrow; Biopsy, Bone Marrow
Procedure: Echocardiography Test — Undergo ECHO
  Other Names: EC; Echocardiography
Procedure: Multigated Acquisition Scan — Undergo MUGA
  Other Names: Blood Pool Scan; Equilibrium Radionuclide Angiography; Gated Blood Pool Imaging; Gated Heart Pool Scan; MUGA; MUGA Scan; Multi-Gated Acquisition Scan; Radionuclide Ventriculogram Scan; Radionuclide Ventriculography; RNV Scan; RNVG; SYMA Scanning; Synchronized Multigated Acquisition Scanning
Drug: UAE Inhibitor TAK-243 — Given IV
  Other Names: AOB87172; MLN7243; TAK-243

SUMMARY:
This phase I trial studies the side effects and best dose of TAK-243 in treating patients with acute myeloid leukemia or myelodysplastic syndromes with increased blasts that has come back (relapsed) or that is not responding to treatment (refractory). TAK-243 may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To establish the recommended phase 2 dose (RP2D) of UAE inhibitor TAK-243 (TAK-243) administered intravenously in a twice-weekly schedule in patients with relapsed/refractory acute myeloid leukemia (AML) or myelodysplastic syndromes (MDS).

SECONDARY OBJECTIVES:

I. To assess the maximum tolerated dose (MTD) evaluated on the first cycle (Day 1 to 21) of TAK-243, its safety profile, and dose limiting toxicities (DLT).

II. To investigate preliminary anti-leukemic activity of TAK-243 monotherapy in patients with AML or MDS.

III. To describe the pharmacokinetic (PK) profile of TAK-243. IV. To describe the pharmacodynamic (PD) effects of TAK-243.

EXPLORATORY OBJECTIVE:

I. To investigate associations between clinical responses and molecular/cytogenetic abnormalities in the leukemia cells or to the PK profile or PD effects of TAK-243.

OUTLINE: This is a dose-escalation study.

Patients receive TAK-243 intravenously (IV) over 30 minutes on days 1, 4, 8, and 11 of each cycle. Cycles repeats every 21 days for up to 12 months in the absence of disease progression or unacceptable toxicity. Patients undergo urine sample collection, bone marrow aspiration and bone marrow biopsy, multigated acquisition scan (MUGA) and echocardiogram (ECHO) during screening and on study, and blood sample collection throughout the trial.

After completion of study treatment, patients are followed up at 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of AML or MDS with increased blasts (MDS-IB) assessed by local laboratory review according to the 2022 World Health Organization (WHO) criteria for myeloid neoplasms. Both patients with MDS-IB1 (5-9% bone marrow blasts) and MDS-IB2 (10-19% bone marrow blasts) are eligible.
* Patients must have relapsed or refractory disease after receiving at least one prior line of therapy
* AML-specific inclusion criteria: Patients with relapsed or refractory AML with >= 5% bone marrow blasts after receiving at least two courses of intensive induction chemotherapy (including, but not limited to, 7+3 regimen, fludarabine, cytarabine, idarubicin and filgrastim [FLAG-Ida] and mitoxantrone, etoposide, and cytarabine [MEC]) or 2 cycles of venetoclax-based lower intensity regimen (azacitidine plus venetoclax or low-dose cytarabine plus venetoclax), and without any other approved therapies available that would be more appropriate in the investigator's judgment. Patients who have received only one course of intensive induction chemotherapy but are not eligible for a second course because of decreased performance status or clear disease progression may be eligible for participation after discussion with the study principal investigator (PI). Patients with concomitant extramedullary disease relapse are eligible to participate, but not patients with isolated extramedullary relapse without bone marrow disease.
* MDS-specific inclusion criteria: Patients with relapsed or refractory MDS-IB with >= 5% bone marrow blasts after at least 4 cycles of hypomethylating agent (HMA)-based therapy or at least two courses of intensive induction chemotherapy and meet criteria for stable disease (SD), progressive disease (PD) or disease relapse according to the International Working Group 2023 response criteria for higher-risk MDS. Patients must not have access to any other approved therapies that would be more appropriate in the investigator's judgment. Patients who have received less than 4 cycles of HMA-based therapy may be eligible to participate after discussion with the study PI if there is clear evidence of progression or intolerance to HMA-based therapy that precludes its continuation.
* Patients must have recovered from the effects of any prior systemic therapy, radiotherapy or surgery:

  * Patients should not have received other investigational therapy within 2 weeks.
  * Patients should not have received standard chemotherapy within 1 week of administration of study drug; hydroxyurea administration (for leukocyte count control) is permitted.
* Age >=18 years. Because no dosing or adverse event data are currently available on the use of TAK-243 in patients <18 years of age, children are excluded from this study.
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2 (Karnofsky >= 50%).
* Serum bilirubin =< 1.5 × institutional upper limit of normal (ULN).

  * Patients with a known history of Gilbert's syndrome may enroll.
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 3 × institutional ULN.
* Serum creatinine < 176 mcmol/L (2 mg/dL) OR
* Creatinine clearance > 60 mL/min based on the Cockcroft-Gault equation.
* Documented normal cardiac function (>= 50%) by echocardiogram or multi-gated acquisition (MUGA) scan.
* HIV-infected patients on effective anti-retroviral therapy with undetectable viral load withing 6 months are eligible for this trial.
* For patients with evidence of chronic hepatitis B virus (HBV) infection, HBV viral load must be undetectable on suppressive therapy if indicated.
* Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load.
* The effects of TAK-243 on the developing human fetus are unknown and ubiquitin-activating enzyme inhibitors are known to be teratogenic. For this reason, female patients must be:

  * Postmenopausal (age-related amenorrhea >= 12 consecutive months or follicle-stimulating hormone > 40 mIU/mL), for at least 1 year before the screening visit, OR
  * Surgically sterile (i.e., who had undergone hysterectomy or bilateral oophorectomy), OR

If they are of childbearing potential:

* Agree to practice 1 highly effective method and 1 additional effective (barrier) method of contraception, at the same time, from the time of signing the informed consent through 4 months after the last dose of study drug (female and male condoms should not be used together), OR
* Agree to practice true abstinence, when this is in line with the preferred and usual lifestyle of the patient. (Periodic abstinence [e.g., calendar, ovulation, symptothermal, postovulation methods] withdrawal, spermicides only, and lactational amenorrhea are not acceptable methods of contraception.) Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.

  * Male patients, even if surgically sterilized (i.e., status post-vasectomy), who:
* Agree to practice effective barrier contraception during the entire study treatment period and through 4 months after the last dose of study drug (female and male condoms should not be used together), OR
* Agree to practice true abstinence, when this is in line with the preferred and usual lifestyle of the subject. (Periodic abstinence [e.g., calendar, ovulation, symptothermal, postovulation methods for the female partner] withdrawal, spermicides only, and lactational amenorrhea are not acceptable methods of contraception.)

  * Ability to understand and the willingness to sign a written informed consent document. Legally authorized representatives may sign and give informed consent on behalf of study participants.
  * Patients should have a minimum life expectancy of 1 month.

Exclusion Criteria:

* Patients with acute promyelocytic leukemia (APL) or AML with t(15;17)(q22;q12) - PML::RARA).
* Patients who have not recovered from adverse events due to prior anti-cancer therapy (i.e., have residual toxicities > grade 1), except anemia, neutropenia or thrombocytopenia of any grade and grade 2 peripheral neuropathy.
* Presence of any other malignancy requiring active therapy.
* Patients who are receiving any other investigational agents.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to TAK-243.
* Concomitant treatment with organic anion transport protein (OATP) and BCRP inhibitors or strong inducers/inhibitors of cytochrome P450 (CYP)3A4/5. Treatment with these agents must be discontinued at least 14 days prior to TAK-243 dosing. Because the lists of these agents are constantly changing, it is important to regularly consult a frequently updated medical reference. As part of the enrollment/informed consent procedures, the patient will be counseled on the risk of interactions with other agents, and what to do if new medications need to be prescribed or if the patient is considering a new over-the-counter medicine or herbal product.
* Presence of an active uncontrolled infection or severe infectious disease, such as severe pneumonia, meningitis, or septicemia.
* Presence of active graft-versus-host disease (GVHD) or continued treatment with systemic immunosuppressive agents following allogeneic hematopoietic stem cell transplantation (HSCT).
* Presence of any co-morbid condition that, in the opinion of the investigator, might compromise the patient's safety, might interfere with participation in the trial or might interfere with the interpretation of trial results.
* Pregnant and lactating/breast-feeding women are excluded from this study because TAK-243 is a UAE-inhibiting agent with the potential for teratogenic or abortifacient effects and there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with TAK-243. Females of child-bearing potential must have a negative serum pregnancy test within 7 days before enrollment and should not be lactating/breast-feeding. Breastfeeding should be discontinued if the mother is treated with TAK-243.
* Major surgery within 14 days before the first dose of any study drug or a scheduled surgery during study period.
* Patients with uncontrolled coagulopathy or bleeding disorder.
* Patients with known hepatic cirrhosis.
* Patients with known active cardiopulmonary disease defined as:

  * Unstable angina withing 3 months prior to first dose of TAK-243;
  * Myocardial infarction (MI) within 6 months prior to first dose of TAK-243 (patients who had MI and/or coronary revascularization more than 6 months before screening and who are without cardiac symptoms may enroll);
  * Congestive heart failure (New York Heart Association [NYHA] Class III or IV;
  * Cardiomyopathy with left ventricular ejection fraction (LVEF) < 50%;
  * Symptomatic pulmonary hypertension.
* Presence of active central nervous system (CNS) involvement (patients with prior CNS leukemia who have negative CNS cytology and who receive periodic prophylactic intrathecal chemotherapy are eligible).
* Patients with clinically significant arrhythmia:

  * History of ventricular fibrillation or torsade de pointes at any time,
  * Episode of grade >= 3 atrial fibrillation or flutter in the last 3 months, defined as symptomatic episode, requiring urgent intervention (cardioversion, pacemaker or ablation) or with life-threatening consequences.
* Uncontrolled high blood pressure (i.e., systolic blood pressure >180 mm Hg, diastolic blood pressure > 95 mm Hg).
* Prolonged rate corrected QT (QTc) interval >= 480 msec, calculated using the Fridericia method.
* Patients with known severe or very severe chronic obstructive pulmonary disease (defined as forced expiratory volume in one second (FEV1) less than 30% or less than 50% of predicted), interstitial lung disease, or pulmonary fibrosis.
* Female patients who intend to donate eggs (ova) during the course of this study or 4 months after receiving their last dose of study drug(s).
* Male patients who intend to donate sperm during the course of this study or 4 months after receiving their last dose of study drug(s).
* Patients with history of neutrophilic dermatosis (e.g. Sweet syndrome, pyoderma gangrenosum), relapsing polychondritis, polyarteritis nodosa and/or giant cell arteritis.
* Patients with VEXAS syndrome (Vacuoles, E1 enzyme, X-linked, Autoinflammatory, Somatic syndrome) or any other autoinflammatory disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2025-03-12 (Actual); Primary Completion 2026-10-24 (Estimated); Study Completion 2026-10-24 (Estimated)

PRIMARY OUTCOMES:
Recommended phase II dose (RP2D) | At 21 days
  RP2D will be identified based on maximum tolerated dose and additional safety data. Primary endpoint will be analyzed on the population assessable for safety of the phase 1 trial (escalation part).

SECONDARY OUTCOMES:
Incidence of adverse events | Up to 30 days after the last dose of TAK-243
  Determined by clinical symptoms/signs, laboratory evaluation and imaging. Graded by Common Terminology Criteria for Adverse Events (CTCAE) version 5.0. Will be recorded in terms of event type, severity, dates of beginning and end, reversibility and evolution. Data will be gathered in tables summarizing toxicities and side effects for each dose level and cycle.
Incidence of serious adverse events | Up to 30 days after the last dose of TAK-243
  Determined by clinical symptoms/signs, laboratory evaluation and imaging. Graded by CTCAE version 5.0. Will be recorded in terms of event type, severity, dates of beginning and end, reversibility and evolution. Data will be gathered in tables summarizing toxicities and side effects for each dose level and cycle.
Incidence of dose-limiting toxicities (DLTs) | Within the first cycle (Up to 21 days)
  DLT will be described in terms of number and incidence rates at each dose level. The number and percentage of patients who will have developed a DLT in each dose level will also be reported.
Rate of complete response (CR) in patients with acute myeloid leukemia (AML) | Up to 1 year
  As defined by European LeukemiaNet criteria. Categorical endpoints (e.g., response) will be reported in terms of counts by dose level.
Rate of complete response with incomplete hematological recovery (CRi), in patients with AML | Up to 1 year
  As defined by European LeukemiaNet criteria. Categorical endpoints (e.g., response) will be reported in terms of counts by dose level.
Rate of CR with partial hematological recovery (CRh) in patients with AML | Up to 1 year
  As defined by European LeukemiaNet criteria. Categorical endpoints (e.g., response) will be reported in terms of counts by dose level.
Rate of partial response (PR) in patients with AML | Up to 1 year
  As defined by European LeukemiaNet criteria. Categorical endpoints (e.g., response) will be reported in terms of counts by dose level.
Rate of morphologic leukemia-free state (MLFS) in patients with AML | Up to 1 year
  As defined by European LeukemiaNet criteria. Categorical endpoints (e.g., response) will be reported in terms of counts by dose level.
Overall response rate (ORR) in patients with AML | Up to 1 year
  Will include CR, CRi plus CRh. Categorical endpoints (e.g., response) will be reported in terms of counts by dose level.
Time to response in patients with AML | From study treatment initiation (Cycle 1 Day 1) to achievement of CR, CRi or CRh, assessed up to
  Categorical endpoints (e.g., response) will be reported in terms of counts by dose level.
Overall survival (OS) in patients with AML | From study treatment initiation to death (of any cause) or last follow-up, assessed at 6 months and 1 year
  OS rates will be reported. OS will be analyzed using the Kaplan-Meier method. The median survival rates will be reported with a 95% confidence interval. Median follow-up will be calculated using the reverse Kaplan-Meier method.
Relapse-free survival (RFS) in patients with AML | From CR, CRi or CRh to the first occurrence of disease relapse, death (of any cause) or last follow-up, whichever occurs first, assessed at 6 months and 1 year
  Will be analyzed using the Kaplan-Meier method. The median survival rates will be reported with a 95% confidence interval. Median follow-up will be calculated using the reverse Kaplan-Meier method.
Rate of CR in patients with myelodysplastic syndrome (MDS) | Up to 1 year
  Categorical endpoints (e.g., response) will be reported in terms of counts by dose level.
Rate of CR equivalent in patients with MDS | Up to 1 year
  Categorical endpoints (e.g., response) will be reported in terms of counts by dose level.
Rate of CR with limited count recovery (CRL) in patients with MDS | Up to 1 year
  Categorical endpoints (e.g., response) will be reported in terms of counts by dose level.
Rate of CR with partial hematologic recovery (CRh) in patients with MDS | Up to 1 year
  Categorical endpoints (e.g., response) will be reported in terms of counts by dose level.
Rate of marrow CR in patients with MDS | Up to 1 year
  Categorical endpoints (e.g., response) will be reported in terms of counts by dose level.
Rate of PR in patients with MDS | Up to 1 year
  Categorical endpoints (e.g., response) will be reported in terms of counts by dose level.
ORR in patients with MDS | Up to 1 year
  Defined by the revised International Working Group 2023 response criteria for higher-risk MDS. Categorical endpoints (e.g., response) will be reported in terms of counts by dose level.
Time to response in patients with MDS | From study treatment initiation (Cycle 1 Day 1) to achievement of CR, CRL or CRh, assessed up to 1 year
  Categorical endpoints (e.g., response) will be reported in terms of counts by dose level.
OS in patients with MDS | From study treatment initiation to death (of any cause) or last follow-up, assessed at 6 months and 1 year
  OS rates will be reported. OS will be analyzed using the Kaplan-Meier method. The median survival rates will be reported with a 95% confidence interval. Median follow-up will be calculated using the reverse Kaplan-Meier method.
Progression-free survival (PFS) in patients with MDS | From study treatment initiation to the first occurrence of progressive disease (PD), relapse from CR (or CR equivalent), death (of any cause), or last follow-up whichever occurs first, assessed at 6 months and 1 year
  PFS rates will be reported. PFS will be analyzed using the Kaplan-Meier method. The median survival rates will be reported with a 95% confidence interval. Median follow-up will be calculated using the reverse Kaplan-Meier method.
Pharmacokinetic measurements | Baseline up to 1 year
  Expressed as area under the curve (AUC), half-life (t1/2), and maximum concentration (Cmax).
Demonstration of UBA1-TAK-243 engagement | Baseline up to 1 year
  Assayed by proprietary monoclonal antibody courtesy of Takeda, to determine target binding and inhibition.
Reductions of protein mono- and poly ubiquitylation | Baseline up to 1 year
  Measured by FK2 antibody. Used as a functional marker of target inhibition.

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume Richard-Carpentier, Principal Investigator — University Health Network Princess Margaret Cancer Center LAO
Locations (4):
- United States (3):
  - Moffitt Cancer Center, Tampa, Florida
  - Northwestern University, Chicago, Illinois
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia
- University Health Network-Princess Margaret Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page
URL: https://grants.nih.gov/policy/sharing.htm